CLINICAL TRIAL: NCT03941691
Title: Chinese Academy of Medical Sciences, Fuwai Hospital
Brief Title: A Trial to Evaluate the Safety and Efficacy of a Fully Degradable Ventricular Septal Defect (VSD) Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Shanghai Shape Memory Alloy Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WQKJJ001
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Ventricular Septal Defect
Keywords: VSD; Ventriculai Septal Defects; amplatzer
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental group is allocated to use novel fully degradable ventricular septal defect closure system manufactured by Shanghai shape memory alloy materials co. LTD.
  Interventions: Device: Fully Absorbable VSD Occlusion System
- Control Group (Active Comparator): Control Group is allocated to use Interposition conveying device for ventricular septal defect closure produced by Shanghai shape memory alloy material co. LTD.
  Interventions: Device: VSD Occluder

INTERVENTIONS:
Device: Fully Absorbable VSD Occlusion System — Under echocardiography guided treatment of VSD with a novel fully degradable clolsure system
  Arms: Treatment Group
Device: VSD Occluder — Under echocardiography guided treatment of VSD with commercially available occluder.
  Arms: Control Group

SUMMARY:
The purpose of this clinical trial is to verify the safety and effectiveness of the Fully Absorbable VSD Occlusion System and VSD Occlusion System produced by Shanghai shape memory alloy materials co., LTD. Clinical trials are designed as prospective, multicenter, randomized controlled, noninferiority clinical trials. Prospective randomized multicenter trial involving about 108 subjects will be enrolled in 4 centers. Patients will be randomized to two groups in equal proportion (54 in each). The success rate of occlusion at 6 months after operation is the main evaluation index in this clinical trial.

DETAILED DESCRIPTION:
1. This is a prospective, multicenter, randomized and noninferiority clinical trial, which is designed to compare the effectiveness and safety with the fully absorbable ventricular septal defect (VSD) occlusion system and VSD occlusion system produced by Shanghai shape memory alloy materials co., LTD.
2. This trial will recruit about 108 subjects from 4 centers. Patients will be randomized to two groups in equal proportion (54 in each). The proposal recruiting period is 12 months and the follow-up will be performed at 1 month, 3 months and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and/or their legal guardians will be informed of the nature of this study and agree to participate in this clinical trial in accordance with all terms of this study.Signed the informed consent approved by the ethics committee, agreed to accept the postoperative treatment program, and completed the follow-up and related examinations as required by the follow-up;
2. Aged from 1 to 60 years old, weight more than 10 kg, male or non-pregnant women;
3. VSD effective shunt ≥3mm, ≤14mm;
4. Distance between the edge of defect and the right aortic valve is more than 3mm, no aortic valve prolapse or moderate aortic regurgitation.

Exclusion Criteria:

1. Irreversible pulmonary vascular disease;Severe pulmonary hypertension with bidirectional shunt;
2. Bleeding disorders or known clotting disorders (including heparin-induced thrombocytopenia),contraindications to antiplatelet therapy, or rejection of transfusions;
3. Sepsis or severe infection within 1 month prior to occlusion;
4. Patients with thrombosis at the occluder placement and venous thrombosis at the catheter insertion site;
5. Cardiac malformation dependent on ventricular septal defect (VSD);
6. Not suitable for treatment with this product.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
success rate of occlusion at 6 months after the surgery | 6 months after the surgery
  Successful occlusion is that when follow-up under echocardiography at 6 months after surgery, the occlusion site shows no residual shunt or only a small amount of residual shunt.

SECONDARY OUTCOMES:
Surgical technique success rate | Immediately after surgery
  After the occluder was implanted with surgical intervention transport device (test group) or occluder and intervention transport device (control group), the occluder was released safely.
technique success rate | Immediately after surgery
  After the occluder was implanted with occluder and surgical intervention transport device (test group) or occluder and intervention transport device (control group), the occluder was released safely and no occluder detachment occurred during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Pan Xiangbin, MD, Ph.D, Principal Investigator — Chinese Academy of Medical Science, Fuwai Hospital
Locations (4):
- China (4):
  - Hefei high-tech cardiovascular hospital, Hefei, Anhui
  - Structral Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality
  - The Second XIANGYA Hospital Of Central South University, Hunan, Changsha
  - Children's Hospital Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03941691/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03941691/ICF_001.pdf